CLINICAL TRIAL: NCT06787183
Title: Efficacy and Safety of Short Course Radiotherapy Combined With CAPOX and PD-1/CTLA-4 Bispecific Antibody QL1706 in Patients With Liver Metastases From Rectal Cancer
Brief Title: SCRT(Short Course Radiotherapy) Combined With CAPOX Plus QL1706 for Rectal Cancer Liver Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCARLET
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Rectal Cancer With Liver Metastases
Keywords: short course radiotheraphy; CAPOX; QL1706 (bifunctional PD1/CTLA4 dual blocker)
MeSH Terms: interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short course radiotherapy combined with CAPOX and QL1706 (Experimental): Two cycles of CAPOX combined with QL1706 were followed by a short course of radiotherapy (CTV 25Gy/5f) and finally two cycles of CAPOX and QL1706.
  Interventions: Radiation: Short course radiotherapy; Drug: Capecitabine; Drug: Oxaliplatin; Drug: QL1706

INTERVENTIONS:
Radiation: Short course radiotherapy — CTV 25Gy/5Fx.
Drug: Capecitabine — 1000mg/m2, d1-14，bid, q3w, 2 cycles.
Drug: Oxaliplatin — 130mg/m2, d1, q3w, 2 cycles
Drug: QL1706 — 5.0 mg/kg, q3w

SUMMARY:
To enhance the treatment efficacy of rectal cancer liver metastasis through a multidisciplinary approach of radiotherapy, immunotherapy, and chemotherapy, and to provide a new direction for the combination treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, any gender.
2. Pathologically confirmed rectal cancer with liver metastases (stage M1).
3. Karnofsky Performance Status ≥70.
4. Adequate organ function, no contraindications to radiotherapy, or immunotherapy.
5. Microsatellite/mismatch repair status MSS/pMMR.
6. No prior chemotherapy or any other anti-tumor treatment before inclusion.
7. No prior immunotherapy.
8. Ability to comply with the study protocol during the study period.
9. Signed written informed consent.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Pathological diagnosis of signet ring cell carcinoma.
3. History of other malignancies within the past 5 years, except cured skin cancer and cervical carcinoma in situ.
4. Uncontrolled epilepsy, central nervous system disorders, or history of psychiatric disorders that, in the opinion of the investigator, may interfere with signing the informed consent form or affect patient compliance with oral medication.
5. Clinically significant (i.e., active) cardiac disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) Class II or greater congestive heart failure, or significant arrhythmias requiring drug intervention (see Appendix 12), or history of myocardial infarction within the past 12 months.
6. Organ transplant recipients requiring immunosuppressive therapy and long-term steroid users.
7. Patients with autoimmune diseases.
8. Severe uncontrolled recurrent infections or other severe uncontrolled comorbidities.
9. Subjects with baseline hematological and biochemical parameters not meeting the following criteria: hemoglobin ≥90g/L; absolute neutrophil count (ANC) .≥1.5×10^9/L; platelets ≥100×10^9/L; ALT, AST ≤2.5 times the upper limit of normal; ALP ≤2.5 times the upper limit of normal; serum total bilirubin <1.5 times the upper limit of normal; serum creatinine <1 times the upper limit of normal; serum albumin ≥30g/L.
10. Known deficiency of dihydropyrimidine dehydrogenase (DPD).
11. Allergy to any investigational drug components.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free-Survival | from enlrollment to 36month

SECONDARY OUTCOMES:
Toxic reaction rate above 3rd degree | from enlrollment to 36month
relapse-free survival | from enlrollment to 36month
overall survival | from enlrollment to 36month

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China